CLINICAL TRIAL: NCT05719389
Title: EFFICACY AND SAFETY OF S.C. INFLIXIMAB IN PATIENTS SWITCHED FROM I.V. FORMULATION OF INFLIXIMAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, GASTROENTEROLOGIST, IRCCS San Raffaele
Other Study IDs: BIO BETTER SWITCH
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases; Rheumatologic Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Collagen Diseases | interventions — CT-P13

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: CT-P13 — CT-P13 is a biosimilar of infliximab approved by EMA since 2015, and it is administered intravenously (i.v.) at a standard dose of 5 mg/kg at week 0, 2, 6 and then every 8 weeks, although the scheduled maintenance regimen can be optimized by administering the drug every 4-6 weeks or increasing the dose up to 10 mg/kg2.The safety profile of CT-P13 SC was comparable to that of CT-P13 i.v.; There were also fewer patients with positive anti-drug antibodies with CT-P13 SC than with CT-P13 i.v.3 At the moment, no data are available on the effectiveness, safety and immunogenicity in a real-world population of patients who have been switched from i.v. to s.c. infliximab.

SUMMARY:
Phase-IV, national, multicentric, non-randomized, observational real-life study. The goal of this stud is to investigate the patient's benefits in terms of quality of life and work ability resulting from the switch from infliximab i.v. to s.c. in patients with gastroenterological or rheumatological indication at month 12.Patients who are eligible but were switched before the inclusion in this study will also be enrolled, and the data already collected according to clinical practice and consistent with the study outcome measures will be used retrospectively. All patients will be followed up according to the standard of care of each participating center.

The main questions it aims to answer are:

1. To investigate the effectiveness at month 2, 6 and 12 after switching to infliximab s.c.
2. To investigate the safety profile at month 2, 6 and 12 after switching to infliximab s.c.
3. To investigate the difference between patients with rheumatological diseases and patients with IBD in terms of quality of life and work, effectiveness and safety at month 2, 6 and 12 after switching.
4. To investigate the presence of baseline predictors for drug persistence at month 12 (sex, age, disease type, disease severity, body mass index, concomitant medications, smoking habit, presence of comorbidities).
5. To investigate whether there is any change between baseline and week 52 in the following aspects:

   * Job type and need for any authorization to go to the hospital to receive the study drug
   * Distance and duration of the travel home-hospital
   * Mode of travel home-hospital
   * Need for a caregiver to be present
   * Time spent at hospital
   * Patient's preference for the way of study drug administration expressed on a 10-grades VAS scale.

The study period for observation will be 12 months from the date of switch. At week 0, month 2, 6 and 12 from the date of the switch, clinical activity, safety data and biomarker levels will be collected.

For those patients who have had an endoscopic evaluation of the disease within 2 months of inclusion and repeat the endoscopic evaluation at 12 months ± 8 weeks, endoscopic data will also be collected (valid only in the presence of IBD).

In those centers where a blood sample to analyze the minimum levels and anti-drug antibodies of infliximab has been collected and/or stored within 2 months prior to the date of transition, the patient will be asked to give informed consent to the use of this sample and to provide a blood sample for the same analysis at week 0, month 2 and 12. These samples will be analyzed and compared to evaluate the immunogenicity of the drug. These analyzes will be centralized in one lab.

DETAILED DESCRIPTION:
250 patients with confirmed diagnosis of Crohn's disease or ulcerative colitis, rheumatoid arthritis, ankylosing spondylitis or psoriatic arthritis;, aged≥ 18, with full ability to understand study procedures and sign an informed consent form, exposed to infliximab i.v. for at least the minimum time required by the current SmPC, and switched to infliximab s.c. 120 mg q2w since the launch date of s.c. infliximab into the Italian market will be prospectively enrolled.

Descriptive analyses will be used for all results. Since there is no control arm, a comparison will be made between the study outcomes and the expected rates reported in the literature for patients treated with infliximab. Survival analyses will be used to acquire and analyze safety and treatment persistence endpoints. Depending on the normality in the distribution of the variables, parametric and non-parametric tests will be used to perform the appropriate statistical analyzes. For all statistical analyzes, a p value <0.05 will be considered as the limit for significance.

Enrollment period:18 months after the approval of the relevant ethical committee Observational period for each patient:12 months from the date of switch

Statistical analysis and publication of results: 6 months after the last patient's follow-up time completion:

Total duration: 3 years

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient of ≥18 years age and no upper age limit
2. Patients with confirmed diagnosis of at least one of the following conditions: Crohn's disease; ulcerative colitis; rheumatoid arthritis4 (2010 ACR/EULAR criteria); ankylosing spondylitis (according to the ASAS modification of the Berlin algorithm for diagnosing ankylosing spondylitis)5; psoriatic arthritis (CASPAR criteria)6.
3. Exposed to i.v. infliximab for at least the minimum time required by the current SmPC, and switched to infliximab s.c. 120 mg q2w prior or at the time of to the inclusion in this study.
4. Treatment with infliximab is according to local approved label
5. Full ability to understand the study procedures and to sign an informed consent form

Exclusion Criteria:

a. Known intolerance/allergy/reaction to infliximab or any excipient included in the s.c. infliximab formulation

1. Non confirmed diagnosis of IBD (unclassified IBD) or not classifiable as having RA or AxSpA or PsA according to the respective criteria
2. Cardiac insufficiency grade IV according to the NYHA scale
3. Active infection at the time of inclusion
4. Pregnancy or lactation at the time of inclusion
5. Active malignancy at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 patients with any indication will be enrolled. Since no previous data are available from the literature, this is a number which is considered reasonable to get adequate magnitude to support the validity of the expected data for the primary outcome.
  At least 10 hospitals across Italy will be involved, where IBD patients and patients with rheumatological disease are regularly followed-up and treated for their condition. The enrollment will be competitive, although all measures will be taken to allow adequate balance in the number of patients enrolled in each center, and in the number of patients with gastroenterological or rheumatological conditions.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with stable or improved from baseline WPAI and SF-36 scores at month 12 s.c. in patients with gastroenterological or rheumatological indication at month 12. | 12 months
  Proportion of patients with stable or improved from baseline WPAI and SF-36 scores at month 12 s.c. in patients with gastroenterological or rheumatological indication at month 12.

SECONDARY OUTCOMES:
Proportion of patients with normal or improved clinical scores at month 2, 6, and 12 | 12 months
  Proportion of patients with normal or improved clinical scores at month 2, 6, and 12
Number, severity, and type of adverse events/ seriuos adverse events through month 12 | 12 months
  Number, severity, and type of adverse events/ seriuos adverse events through month 12
f) Difference between patients with rheumatological diseases and patients with IBD in terms of quality of life and work, effectiveness and safety at month 2, 6 and 12 after switching | 12 months
  f) Difference between patients with rheumatological diseases and patients with IBD in terms of quality of life and work, effectiveness and safety at month 2, 6 and 12 after switching

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Irccs Ospedale San Raffaele, Milan, Italy